CLINICAL TRIAL: NCT06405243
Title: The Combination of Myoinositol, L-arginine and Chromium With Letrozole for Ovulation Induction in Polycystic Ovarian Syndrome Patients
Brief Title: Myoinositol, L-arginine and Chromium With Letrozole for Ovulation Induction in Polycystic Ovarian Syndrome Patients
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Sara Abdallah Mohamed Salem, principle investigator/Lecturer of Gynecology and obstetrics Faculty of medicine Beni-Suef University, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: myoinositol/letrazol/pco
Record Dates: First submitted 2024-05-04; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic Ovary Syndrome; letrazole; myoinositol; L-arginine; Chromium
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Inositol; Chromium; Arginine; Letrozole

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- myoinositol (Experimental): patients will be treated for 12 weeks myoinositol (2gm /day) with ovulation induction by letrazole regimen for 3 consecutive cycl
  Interventions: Drug: Myoinositol; Drug: Letrozole 2.5mg
- chromium (Experimental): patients will be treated for 12 weeks chromium ( 281.569 mcg/ day) with ovulation induction by letrazole regimen for 3 consecutive cycles
  Interventions: Drug: Chromium; Drug: Letrozole 2.5mg
- L-arginine (Experimental): : patients will be treated for 12 weeks with L-arginine (500 mg once daily in the morning) with ovulation induction by letrazole regimen for 3 consecutive cycles.
  Interventions: Drug: l-arginine; Drug: Letrozole 2.5mg

INTERVENTIONS:
Drug: Myoinositol — Myoinositol decreases insulin resistance and consequently increased intracellular glucose uptake, restore the metabolic profile and induce ovulation in PCOS patients with infertility, in addition to its good safety profile
  Other Names: femtonex
  Arms: myoinositol
Drug: Chromium — chromium picolinate may potentiates the therapeutic effect of letrozol on pituitary hormones (FSH and LH), improvement of ovulation, normalization of Estrogen level, improvement of endometrial thickness related to ovulation
  Other Names: chromax
  Arms: chromium
Drug: l-arginine — new antioxidant that minimizes the inflammatory reaction, the hormonal imbalance, and the metabolic disturbances in PCO
  Other Names: Blue ox
  Arms: L-arginine
Drug: Letrozole 2.5mg — selective aromatase inhibitor
  Other Names: femara

SUMMARY:
The aim of the study is to compare and assess the efficacy of combined letrozole with myoinositol, chromium, or L-arginine in infertile women with PCOS. This study will help in the investigation of alternative therapeutic modalities for fertility improvement in polycystic ovarian syndrome

DETAILED DESCRIPTION:
d prospective Study Trial. We will recruit patients diagnosed with PCOS according to Rotterdam criteria of PCOS and who present to outpatient clinics at Beni-Suef University Hospital. Infertile women will be randomized to receive letrozole (2.5 mg for 5 days from 3rd day of patients' menstrual cycle) combination with myoinositol, chromium or L-arginine

ELIGIBILITY:
Inclusion Criteria:

* Primary or secondary infertility associated with PCOS as defined by the revised Rotterdam criteria
* Normal values of the following laboratory tests: thyroid function, prolactin level, and husband's sperm analysis and hysterosalpingography

Exclusion Criteria:

1. Patients with a history of systemic diseases such as liver, kidney, cardiovascular, diabetes (type I or II) or malignancy.
2. Patients who consumed myoinositol, metformin, SGLT2 or drugs effecting insulin secretion or clomiphene citrate in the previous 2 months.

3. Use of hormonal medications, lipid-lowering agents (statins, etc.), anti-obesity drugs or medications for weight loss in the previous 2 months.

4. Patients with hormonal disorders such as hyperprolactinemia, hypo or hyperthyroidism or Cushing syndrome. 5. Presence of hypersensitivity to any of the study medications.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-06-30 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
ovulation | 3 cycles ( 3 months / one month for each cycle)
  trans-vaginal ultrasound shows dominant follicle more than 18mm

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Beni-suef university Hospital, Banī Suwayf
  - Beni-suef university, Banī Suwayf

IPD SHARING:
Plan to Share IPD: No